CLINICAL TRIAL: NCT03073083
Title: Graft Selection in Anatomic Anterior Cruciate Ligament Reconstruction: Patella, Hamstrings or Quadriceps Tendon Autograft
Brief Title: Graft Selection in Anatomic Anterior Cruciate Ligament Reconstruction
Acronym: Grafttype
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedisch Centrum Oost Nederland (Other)
Collaborators: Martini Hospital Groningen (Other); Gelderse Vallei Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL52749.044.16
Record Dates: First submitted 2017-02-23; First posted 2017-03-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: autograft
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hamstring tendon autograft (Active Comparator): ACL reconstruction surgery with hamstring tendon autograft
  Interventions: Procedure: Hamstring tendon autograft
- Patella tendon autograft (Active Comparator): ACL reconstruction surgery with pattella tendon autograft
  Interventions: Procedure: Pattella tendon autograft
- Quadriceps tendon autograft (Active Comparator): ACL reconstruction surgery with quadriceps tendon autograft
  Interventions: Procedure: Quadriceps tendon autograft

INTERVENTIONS:
Procedure: Hamstring tendon autograft — ACL reconstruction surgery with hamstring tendon
  Other Names: all-inside AMPS technique Arthrex
  Arms: Hamstring tendon autograft
Procedure: Pattella tendon autograft — ACL reconstruction surgery with patella tendon
  Other Names: Smith and Nephew
  Arms: Patella tendon autograft
Procedure: Quadriceps tendon autograft — ACL reconstruction surgery with quadriceps tendon
  Other Names: all-inside AMPS technique Arthrex
  Arms: Quadriceps tendon autograft

SUMMARY:
A rupture of the anterior cruciate ligament (ACL) is a severe injury of the knee. The current gold Standard treatment for young and active patients with instability, is a surgical ACL reconstruction. However, there still is no consensus on which graft is best suited for this.The aim of the current multi-center randomized controlled trial was to investigate the hypothesis that an anatomic single bundle anterior cruciate ligament reconstruction with a (flat) quadriceps tendon autograft is at least as effective as reconstruction of the ruptured anterior cruciate ligament with a patella tendon autograft or a hamstringtendon autograft, in terms of failure, measured 2 years postoperatively. Failure is defined gedefinieerd as pathologicai laxity, complaints of knee instability in the absence of any pathological laxity and/or discontinuïty ofthe graft on MRl or arthroscopy.

DETAILED DESCRIPTION:
A rupture of the anterior cruciate ligament (ACL) is a severe injury of the knee. The current gold Standard treatment for young and active patients with instability, is a surgical ACL reconstruction. However, there still is no consensus on which graft is best suited for this.

Paradigms on the different types of auto grafts and their weaknesses and benefits originate mostly from the eighties and nineties, when the patella tendon was being replaced by the hamstring graft as the 'new' gold standerd. Nowadays, the philosophy of isometrie tunnel placement has been abandoned, and has been replaced by the philosophy of anatomie reconstructions. The question then arises: Are the results of the comparative studies, and the current paradigms, still applicable, now that the philosophy has transitioned from isometric to anatomic tunnel placement? Irrespective of the disadvantages compared to the patellatendon autograft, such as a higher re-rupture and revision percentage when used in patients under 25 years old, the hamstring autograft is currently the most used graft for ACL reconstruction worldwide. The question then arises: is it justified that the hamstringgraft is the most used graft worldwide? Rehabilitation protocols are often not, or poorly, described, despite it's significant effect on the outcome and co morbidity of an ACL reconstruction. Especially anterior knee pain, which is often mentioned as a disadvantage of the patellagraft, is significantly influenced by rehabilitation protocols. The introduction and implementation of a nation-wide evidence-based rehabilitation protocol in The Netherlands created uniformity of rehabilitation treatment, and the possibility to generalize scientific conclusions. The question then arises: Due to new insights in rehabilitation and implementation of new protocols, is the anterior knee pain, the often mentioned disadvantage ofthe patelia tendon graft, stiil a relevant disadvantage? The quadriceps tendon autograft is a less often used graft. Nevertheless, research has shown that it seems like a good alternative for the patella tendon and hamstring autograft. Functional outcome is similar, while less donorsite morbidity is reported compared to the patellatendon and hamstring autograft. The question then arises: Is it fair that the quadriceps tendon is rarely used as an autograft for ACL reconstruction? Increasing knowledge of the anatomy of the ACL results in new insights in the methods to achieve true anatomie ACL reconstruction. New arguments support the use of the patella tendon - and even the quadriceps tendon - over the use of the hamstringgraft, because their anatomic similarities to the anterior cruciate ligament might be better suited to restore knee kinematics. The question then arises: are the flat-shaped patella tendon autograft and quadriceps tendon autograft better suited to restore the anatomy of the ruptured ACL than the round hamstring graft? Hypothesis Tlie hypothesis is that anatomic reconstruction ofthe ruptured anterior cruciate ligament with a (flat) quadriceps tendon autograft is at least as effective as reconstruction of the ruptured anterior cruciate ligament with a patella tendon autograft or a hamstring tendon autograft, in terms of failure, measured 2 years postoperatively. Failure is defined as pathological laxity, complaints of knee instability in the absence of any pathological laxity and/or discontinuïty of the graft on MRl or arthroscopy.

Objective of the study:

Primary objective:

To investigate the hypothesis that an anatomic single bundle anterior cruciate ligament reconstruction with a (flat) quadriceps tendon autograft is at least as effective as reconstruction of the ruptured anterior cruciate ligament with a patella tendon autograft or a hamstring tendon autograft, in terms of failure, measured 2 years postoperatively. Failure is defined gedefinieerd as pathologicai laxity, complaints of knee instability in the absence of any pathological laxity and/or discontinuïty of the graft on MRl or arthroscopy.

**Graft failure at 2 years (originally registered). Due to premature termination, this outcome was underpowered and analyzed exploratorily. The IKDC Subjective Knee Form score was analyzed as the main outcome in the final report.**

Secondary objectives:

patiënt reported outcome measures (PROMs), clinimetrics, radiological assessment, duration of rehabilitation necessary for return to sports and daily activities and the level of sport activities to which the patiënt returned, in patients treated with an anterior cruciate ligament reconstruction using a patellatendon autograft, hamstringtendon autograft of quadricepstendon autograft, as measured in the short-term (6 weeks, 6,9,12 months postoperatively), mid-term (2 years postoperatively) and long-term (5 and 10 years postoperatively).

Study design:

Multicenter blocked stratified randomised controlled trial with varying block sizes (n=3, 6, 9, 12). Patients with an anterior cruciate ligament rupture, confirmed by an orthopaedie surgeon (as evident from anamnesis, physical examination and radiographic imaging) who meet the inclusion criteria and do not have any of the exclusion criteria, will be asked to partieipate in this study.

Baseline measurements will be performed, after informed consent is obtained. Allocation of treatment of the included patients will be performed in the operating room (OR), where patients will be randomised (blocked and stratified) per clinic, to have ACL reconstruction with a patella tendon autograft, hamstring tendon autograft or quadriceps tendon autograft. Stratification will be based on age (18-25 and >25), level of sport activities (Tegner Activity Level Scale 5-7 and 8-10) and surgeon.

Follow-up identical to the follow-up of standard care, with standard checkups after 6 weeks, 6, 9, months and 1 and 2 years. Two extra follow-up moments (after 5 and 10 years) will be planned.

** Study inclusion stopped early due to slower-than-expected recruitment (patient preference, COVID-19) and changes in standard care including the addition of a Lemaire procedure. Continuing without it was no longer appropriate. The achieved sample size allowed adequate power (80%) for non-inferiority analysis of the IKDC subjective score (-10 points difference, n = 23 per group). Follow-up of enrolled participants continues.**

ELIGIBILITY:
Inclusion Criteria:

* Patients active in sports, Tegner =/>5
* Primary ACL rupture, evident from anamnesis (acute trauma, snapping sensation, swelling within several hours, feeling of instability), physical examination (positive Lachman test, anterior drawertest and/or pivot shift test), radiograph and MRl
* Willing to comply to the suggested (nationwide standard) rehabilitation protocol, supen/ised by a NFVS registerd sport-physical therapist
* <6 months between initial trauma and surgery

Exclusion Criteria:

* History of knee surgery on the same side
* History of tendon removal on the same side
* Accompanying ligament injury ofthe knee, evident from anamnesis, physical examination, radiograph and MRl, defined as an ACL rupture in combination with a posterior cruciate ligament or collateral ligament injury,
* Peroperative discovery of cartilage damage; larger than 2cm2 and more than 50% depth
* Peroperative discovery of meniscus injury witch requires a meniscectomy of more than 20% or meniscus sutures
* Osteoarthritis of Kellgren and Lawrence grade 2 or more, as evident from the radiograph
* Severe malalignment of the leg
* Tendency to form excessive scar tissue, such as arthrofibrosis
* Muscular, neurological or vascular anomalies that influence healingtime or rehabilitation
* Infection
* Known hypersensitivity to any of the used materials
* Long term relevant medication use such as prednisolone or cytostatics
* Pregnancy at the time of inclusion or surgery
* Known osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Physical examination ACL Failure | 2 years after ACL reconstruction surgery
  Presence / absence of anterior cruciate ligament failure. Failure is defined as pathologicai laxity, complaints of knee instability in the absence of any pathological laxity and/or discontinuïty ofthe graft on MRl or arthroscopy.
  Graft failure at 2 years (originally registered). Due to premature termination, this outcome was underpowered and analyzed exploratorily. The IKDC Subjective Knee Form score was analyzed as the main outcome in the final report. The IKDC subjective score was already powered at study design (-10 points non-inferiority margin; n = 23 per group, 80% power).

SECONDARY OUTCOMES:
quality of life (ACL-QoL) | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  level of self-reported quality of life
functional knee and health status (IKDC) | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  level of functional knee and current health status
physical examination of knee (in)stability | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  instability in the absence of any pathological laxity and/or discontinuïty of the graft on MRl or arthroscopy.
Knee and Injury Osetoarthritis Outcome Score questionnaire (KOOS) | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  self-reported level of physical activity in daily life
sports intensity questionnaire (Tegner Activity Level) | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  self-reported level of pivoting sports execution
questionnaire | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  level of physical activity (Lysholm score)
knee pain | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  self-reported level of pain during activity and rest on visual analogue scale
Instability knee | preoperative, 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  VAS score (patient perception)
satisfaction with result of ACL surgery | 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  self-reported level of satisfaction with ACL surgery on visual analogue scale
physical examination | 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  degree of knee (in)stability during jumping tests (Leg Symmetry Index)
physical examination | preoperative, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  degree of knee (in)stability in strenght (Leg Symmetry Index)
Lachman test | 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  physical examination: degree of knee (in)stability measured by rollimeter (operated-nonoperated side ratio)
Degree of Osteoarthritis on x-ray | Baseline, 1,2,5 10 years after ACL reconstruction surgery
  Kellgren-Lawrence classification will be applied to assess the degree of osteoarthritis

OTHER OUTCOMES:
Knee instability during jumping movements | 1 and 2 years after ACL reconstruction surgery
  Measured during jumping test. At OCON patients will be equiped with 3D accelerometer sensors in order to quantify the degree of (in)stability of the affected knee during the execution of jump tests under the supervision of a specialized sports physiotherapist
Complications and other adverse events | 6 wks, 6 months, 9 months, 1, 2, 5 10 years after ACL reconstruction surgery
  number and type complications and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: R.A.G Hoogeslag, MD, Principal Investigator — OCON
Locations (2):
- Netherlands (2):
  - Martini Hospital Groningen, Groningen
  - OCON, Hengelo

IPD SHARING:
Plan to Share IPD: No